CLINICAL TRIAL: NCT03833869
Title: The Effect of Assisted Hatching on Implantation Rate in Frozen Blastocyst Transfer - a Prospective Randomized Controlled Study
Brief Title: Assisted Hatching in Frozen Blastocysts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Hadas Ganer Herman, Principal Investigator, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0020-19-WOMC
Record Dates: First submitted 2019-02-06; First posted 2019-02-07 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-02

CONDITIONS: ART

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assisted hatching (Experimental): Five-day frozen embryos will undergo assisted hatching prior to embryo transfer
  Interventions: Procedure: Assisted hatching
- Control (No Intervention): Five-day frozen embryos will not undergo any additional procedures prior to embryo transfer

INTERVENTIONS:
Procedure: Assisted hatching — Controlled hatching of the zona pellucida in the laboratory prior to embryo transfer
  Arms: Assisted hatching

SUMMARY:
The current study aims to assess the effect of assisted hatching on the implantation rate of frozen blastocytes.

DETAILED DESCRIPTION:
The Zona Pellucida protects the ovum from the penetration of multiple sperm, and from mechanical and physiological damage until the fertilized ovum reaches the uterus. Subsequently, spontaneous hatching occurs, and enables the embryo to attach to the endometrium. The technique of assisted hatching was originally investigated as a means to improve implantation in cases of zona hardening, and is commonly performed in 3-day embryos. In the current study, the investigators aim to investigate the effect of assisted hatching on 5-day frozen embryos.

ELIGIBILITY:
Inclusion Criteria:

* In-vitro fertilization patients at the investigators' institution, intended to undergo a transfer of a frozen five-day embryo (blastocyte)
* 18 to 39 years old
* First to third treatment cycle
* Patient has previously had a maximum of four embryos transferred.

Exclusion Criteria:

* Over 40 years old
* Congenital or acquired uterine malformations
* Hydrosalpinx
* Chronic autoimmune diseases
* Embryo intended to be undergo preimplantation genetic diagnosis

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Implantation rate | Five to six weeks following embryo transfer
  Number of gestational sacs demonstrated on ultrasound divided by the number of embryos transferred (expressed as percentage)

SECONDARY OUTCOMES:
Chemical pregnancy | Five to six weeks following embryo transfer
  Increase and subsequent decrease in beta HCG levels with no evidence of gestational sac on ultrasound
Early spontaneous abortion | Up to 15 weeks from embryo transfer
  Spontaneous abortion of pregnancy during the first trimester of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Hadas Ganer Herman, MD, Principal Investigator — Edith Wolfson Medical Center
Locations (1):
- Edith Wolfson Medical Center, Holon, Israel